CLINICAL TRIAL: NCT05182463
Title: Real World Study of Peginterferon Alpha-2b Treatment for Inactive Chronic Hepatitis B Patients: E-Cure Study
Brief Title: Peginterferon Treatment Study for Inactive Chronic Hepatitis B Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, Director of the infectious diseases department, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2021]02-373-01
Record Dates: First submitted 2021-12-18; First posted 2022-01-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B, Chronic
Keywords: inactive chronic hepatitis B; functional cure
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b; Nucleosides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Sequential Combination Group (Experimental): Oral nucleos(t)ide analogues (NAs) (Entecavir(ETV), Tenofovir disoproxil fumarate tablets(TDF) or Tenofovir Alafenamide Fumarate(TAF)) is used for 12-24 weeks, followed by combination therapy with peginterferon α-2b. The Maximum course is 96 weeks. Follow-up period is 144 weeks.
  Interventions: Drug: Peginterferon Alfa-2B; Drug: Nucleoside Analogs
- Initial Combination Group (Experimental): NAs combined with peginterferon are used for 12-24 weeks, followed by peginterferon α-2b. The Maximum course is 96 weeks. Follow-up period is 144 weeks.
  Interventions: Drug: Peginterferon Alfa-2B; Drug: Nucleoside Analogs
- Whole-course Combination Group (Experimental): NAs combined with peginterferon are used for a maximum course of 96 weeks. Follow-up period is 144 weeks.
  Interventions: Drug: Peginterferon Alfa-2B; Drug: Nucleoside Analogs
- Peginterferon Monotherapy Group (Experimental): Peginterferon is used for a maximum course of 96 weeks. Follow-up period is 144 weeks.
  Interventions: Drug: Peginterferon Alfa-2B
- NAs Monotherapy Group (Experimental): NAs is used for a maximum course of 96 weeks. Follow-up period is 144 weeks.
  Interventions: Drug: Nucleoside Analogs

INTERVENTIONS:
Drug: Peginterferon Alfa-2B — Different usage of peginterferon Alfa-2B and/or Nucleos(t)ide analogs in arm/group descriptions are depended on the wishes of the patient and the advice of the attending doctor.
  Arms: Initial Combination Group; Peginterferon Monotherapy Group; Sequential Combination Group; Whole-course Combination Group
Drug: Nucleoside Analogs — Nucleos(t)ide analogs refer to one of the first-line drugs, including ETV, TDF and TAF.
  Arms: Initial Combination Group; NAs Monotherapy Group; Sequential Combination Group; Whole-course Combination Group

SUMMARY:
There are about 400 million chronic hepatitis B virus (HBV) infection patients worldwide, posing a serious threat to global public health security. In China, HBV infection occured mainly in the perinatal period or infants, and about 10% of patients in the immune tolerance stage spontaneously transit to the immune clearance stage every year and become HBeAg-negative chronic HBV infection, resulting in a significant increase in the number of inactive chronic hepatitis B (CHB) patients.

In recent years, different guidelines have not reached consensus on the need to initiate antiviral therapy for inactive CHB patients: In the guidelines of Asian Pacific Association for The Study of Liver(APASL)-2015 and American Association for the Study of Liver Diseases(AASLD)-2018, antiviral therapy is generally not recommended for this group of patients, and regular outpatient follow-up is recommended. Guideline of European Association for the Study of the Liver(EASL)-2017 suggests that people with a family history of cirrhosis and liver cancer at this stage could be treated with antiviral therapy even if they did not meet the indications of antiviral therapy. According to Guidelines for the Prevention and Treatment of Chronic Hepatitis B (version 2019) of China, antiviral therapy is still recommended for some patients with inactive HBsAg carrier status who are HBV DNA positive and meet the treatment indications. Studies have shown that some patients in immune tolerance stage may enter the immune clearance stage and have hepatitis flare. Patients of inactive CHB have the potential to develop HBeAg-negative CHB, and studies of long-term follow-up in this population have indicated the risk of hepatocellular carcinoma. With the popularization of the concept of functional cure for chronic hepatitis B, more and more people with inactive CHB have a strong desire for treatment. In recent years, several studies have demonstrated that Pegylated-interferon therapy can achieve high functional cure rate in patients with inactive CHB.

The purpose of this study is to establish a national multi-center, prospective real world study to compare the efficacy of different antiviral treatment regimens for patients with inactive CHB and seek for the factors of functional cure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60, no gender limitation
* HBsAg is positive for more than 6 months
* Hepatitis B e antigen(HBeAg) is negative and anti-HBe is positive
* Serum HBV DNA is less than 2000 IU/mL
* Alanine aminotransferase(ALT) and/or Aspartate aminotransferase(AST) is normal
* No antiviral durg (including nucleos(t)ide analogue and interferon) was used before enrollment
* Good compliance and voluntarily signed informed consent

Exclusion Criteria:

* Allergic to pegylated interferon α-2b
* Any indication of liver cirrhosis
* Coinfection with hepatitis A virus(HAV), hepatitis C virus(HCV), hepatitis D virus(HDV), hepatitis E virus(HEV) or human immunodeficiency virus(HIV)
* Combined with other liver diseases (including drug-related, alcoholic, autoimmune, genetic metabolic liver diseases, etc.)
* There are serious lesions in the important organs, such as heart, lung, kidney, brain and fundus
* Patients with autoimmune diseases, unstable diabetes or thyroid diseases(hyperthyroidism or hypothyroidism)
* Confirmed or suspected liver cancer or other malignant tumors
* Patients after or preparing for organ transplantation
* Peripheral blood white blood cell count < 3.5×109/L and/or platelet count < 80×109/L
* Under immunosuppressant treatment
* Pregnant or planned pregnancy in a short term or lactation patients
* Alcohol abuse (average alcohol intake is more than 40 g/d in males or 20g/d in women) or drug addicts
* Present or past history of mental or psychological diseases
* Other conditions that the investigators deem inappropriate for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-08 (Actual); Primary Completion 2026-12-13 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
HBsAg clearance rate | From date of the beginning of treatment until the date of the end of treatment, assessed up to 96 weeks
  HBsAg is detected by Roche or Abbott productions, of which the lower limit is 0.05 IU/ml

SECONDARY OUTCOMES:
HBsAg serological conversion rate | From date of the beginning of treatment until the date of the end of treatment, assessed up to 96 weeks
  HBsAg is detected by Roche or Abbott productions, of which the lower limit is 0.05 IU/ml
The magnitude of HBsAg decline from baseline | through treatment completion, an anticipated period of 96 weeks
  HBsAg is detected by quantitative assays from Roche or Abbott
The magnitude of HBV-DNA decline from baseline and the undetectable rate | through treatment completion, an anticipated period of 96 weeks
  HBV-DNA is detected by assays from Roche or Abbott, of which the lower limit is 15 or 10 IU/ml.
HBsAg clearance rate, HBsAg serological conversion rate and maintenance response rate of HBsAg clearance | through follow-up completion, an anticipated period of 144 weeks
  HBsAg is detected by Roche or Abbott productions, of which the lower limit is 0.05 IU/ml

CONTACTS AND LOCATIONS:
Overall Officials: Zhiliang Gao, Doctor, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University; Guizhou Zou, Principal Investigator — The Second Hospital of Anhui Medical University; Jiabin Li, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Zhende Lin, Principal Investigator — Anxi County Hospital; Guoxin Hu, Principal Investigator — SHENZHEN HOSPITAL of PEKING UNIVERSITY; Youping Lin, Principal Investigator — Dongguan Binhai Bay Central Hospital; Sichun Yin, Principal Investigator — Dongguan Ninth People's Hospital; Songmei He, Principal Investigator — Dongguan People's Hospital; Zengjia Xu, Principal Investigator — Dongyuan People's Hospital; Hui Shen, Principal Investigator — DuShanZi People's Hospital; Haifei Luo, Principal Investigator — First People's Hospital of Foshan; Wenhua Zhang, Principal Investigator — Gansu Wuwei Tumor Hospital; Maosheng Wu, Principal Investigator — Guangdong Second Provincial People's Hospital; Dong Wei, Principal Investigator — Guangzhou Second traditional Chinese Medicine hospital; Wenli Chen, Principal Investigator — Guangdong Provincial People's Hospital; Bihua Gao, Principal Investigator — Beihai People's hospital; Guifang Tang, Principal Investigator — Nanxishan Hospital of Giang xi zhuang Autonomous Region; Huaiyu Song, Principal Investigator — THE PEOPLE'S HOSPITAL OF GUANGXI ZHUANG AUTCNOMOUS REGION; Zhuxiang Zhao, Principal Investigator — The First Municipal Hospital of Guangzhou; Xihua Fu, Principal Investigator — Guangzhou Panyu Central Hospital; Runqi Luo, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University; Shi Ouyang, Principal Investigator — Fifth Affiliated Hospital of Guangzhou Medical University; Chunlan Zhang, Principal Investigator — GUANGZHOU EIGHTH PEOPLE'S HOSPITAL GUANGZHOU MEDICAL UNIVERSITY; Riying Lv, Principal Investigator — Guigang city People's Hospital; Bigang Xiong, Principal Investigator — GuiYang Public Health Clinlcal Center; Hong Peng, Principal Investigator — the People's Hospital of Guizhou; Sufen Zhou, Principal Investigator — The First Affiliated Hospital of Guizhou University of Traditional Chinese Medicine; Quan Zhang, Principal Investigator — The Affiliated Hospital Of Guizhou Medical University; YongChao Xian, Principal Investigator — The Third People's Hospital of Guilin; Ganwen Li, Principal Investigator — The Third Affiliated Hospital of Sun Yat-Sen Unlversity Yuedong hospital; Jinyu Xia, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University; Bihui Zhong, Principal Investigator — The First Afiliated Hospital Sun Yat-sen University; Minhui Xiao, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Wenjun Gao, Principal Investigator — Zhongshan Sencond People's Hospital; Gang Li, Principal Investigator — The fourth people's Hospital of Zibo; Yangwen Luo, Principal Investigator — Zunyi Medical College; Jie Chen, Principal Investigator — The Second People's Hospital OF YULIN; Xiaochao Qin, Principal Investigator — Red Cross Hospital of Yulin City; Wuhai Qin, Principal Investigator — teaditional chinese medicine hospital of YULIN; Hongshun Fan, Principal Investigator — Yuebei Second People's Hospital; Ming Jiang, Principal Investigator — Guilin Municipal Hospital of Traditonal; Feng Lin, Principal Investigator — HANNAN GENERAL HOSPITAL; Chengfang Zheng, Principal Investigator — Hainan Western Central Hospital; Zhentao Gu, Principal Investigator — Heyuan people's Hospital; Fan Li, Principal Investigator — THE PEOPLE'S HOSPITAL of HEZHOU; Qin Yan, Principal Investigator — Huazhong University of Science and Technology Union Shenzhen Hospital; Zhanzhou Lin, Principal Investigator — Huizhou Municipal Central Hospital; Hui Chen, Principal Investigator — Hepatobiliary Hospital Of JiLin; Xujing Liang, Principal Investigator — First Affiliated Hospital of Jinan University; Bin Liu, Principal Investigator — The Affiliated Shunde Hospital of Jinan University; Changzheng Hu, Principal Investigator — Jiangmen Central Hospital; Xingchuan Wang, Principal Investigator — The 924th Hospital of the PLA joint Logistic support Force; Chengzu Lin, Principal Investigator — Jinjiang City Hospital; Guihua Su, Principal Investigator — the First People's Hopistal of Kashi; Yi Wang, Principal Investigator — Karamay Central Hospital of Xinjiang; Yuqin Xu, Principal Investigator — The 962th Hospital of the PLA joint Logistic support Force; Lingyi Zhang, Principal Investigator — Lanzhou University Second Hospital; Xiaorong Mao, Principal Investigator — LanZhou University; Hong Wan, Principal Investigator — Lanzhou University Second Hospital; Qian Guo, Principal Investigator — LIU ZHOU WORKER'S HOSPITAL; Liu He, Principal Investigator — LIU ZHOU PEOPLE'S HOSPITAL; Zhengxiao Zhao, Principal Investigator — LIU ZHOU TRADITIONAL CHINESE MEDICAL HOSPITAL; Yan Lincan, Principal Investigator — Long yan hospital of traditional Chinese medicine; Feng Min, Principal Investigator — army 73rd group military hospital; Xiqiu Zeng, Principal Investigator — Mudanjiang Kangan Hospital; Shuilin Sun, Principal Investigator — Second Affiliated Hospital of Nanchang University; Xiaoping Wu, Principal Investigator — The First Affiliated Hospital of Nanchang University; Keqin Zhang, Principal Investigator — The Ninth Hospital of Nanchang; Hong Li, Principal Investigator — Southern Medical University, China; Jianzhen Yao, Principal Investigator — Putian Hanjiang Hospital; Liqin Cai, Principal Investigator — The First Hospital of Putian City; Rongxian Qiu, Principal Investigator — The Affiliated Hospital of Putian University; Sandu Liu, Principal Investigator — The People's Hospital Of QianNan; Qinghua Lu, Principal Investigator — The Fourth People's Hospital of Qinghai Province; Ying Deng, Principal Investigator — The Sixth Affiliated Hospital of Guangzhou Medical University; Xingnan Pan, Principal Investigator — Quanzhou Decheng hospital; Ruyi Guo, Principal Investigator — Quanzhou First Hospital; Wenke Li, Principal Investigator — Quanzhou Hospital of traditional Chinese Medicine; Huiwen Song, Principal Investigator — SanMing First Hospital; Xiulan Xue, Principal Investigator — The First Affiliated Hospital of Xiamen University; Qianguo Mao, Principal Investigator — Xiamen Hospital of Traditional Chinese Medicine; Haidong Zhao, Principal Investigator — Xiamen Chang gung hospital; Yanhui Zu, Principal Investigator — Shan dong public Health Clinical Center; Ruilie Chen, Principal Investigator — Shantou Central Hospital; Shu Yang, Principal Investigator — Shenzhen Bao'an People's Hospital; Jun Chen, Principal Investigator — Shenzhen Third People's Hospital; Yanyao Yin, Principal Investigator — Shenzhen Luohu Hospitai of Traditional Chinese Medicine; Rongshan Fan, Principal Investigator — Shenzhen Hospital of Integrated Traditional Chinese and Western Medicine; Guangdong Tong, Principal Investigator — SHEN ZHEN TRADITIONAL CHINESE MEDICINE HOSPITAL; Weize Zuo, Principal Investigator — The First Affiliated Hospital of Shihezi University School of Medicine; Bin Zhou, Principal Investigator — Weihai Chest Hospital; Huanwei Zheng, Principal Investigator — Shijiazhuang Hospital of Traditional Chinese Medicine; Chuantiao Zhang, Principal Investigator — Shishi General Hospital; Qing Ye, Principal Investigator — Tianjin Third Central Hospital; Xin Chen, Principal Investigator — Tianjin First Hospital; Changxia Niu, Principal Investigator — Tianshui First people's hospital; Jiancheng Zhang, Principal Investigator — Tianshui traditional Chinese medicine hospital; Ruihai Zhu, Principal Investigator — Weifang People's Hospital; Zhushi Liang, Principal Investigator — The Third People's Hospital of Wuzhou; Qingming Zheng, Principal Investigator — Fujian Xianyou General Hospital; Xiaobo Lu, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Xiaozhong Wang, Principal Investigator — Traditional Chinese Medicine Hospital of Xinjiang; Huanwen Chen, Principal Investigator — XING AN COUNTY PEOPLE'S HOSPITSL; Haifeng Yu, Principal Investigator — YANTAI QISHAN HOSPITAL; Shengtao Zeng, Principal Investigator — Yili Prefecture Infectious Disease Hospital; Lei Li, Principal Investigator — Anhui Provincial Hospital; Weibing Shi, Principal Investigator — The First Affiliated Hospital of Anhui University of Chinese Medicine; Chuanmiao Liu, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Mei Cai, Principal Investigator — Cangzhou Third Hospital; Lijuan Guan, Principal Investigator — The 2nd Hospital of da qing City; Riwang Hu, Principal Investigator — The 4th People's Hospital of da tong city; Jianli Huang, Principal Investigator — Yongchun County Hospital; Yueyong Zhu, Principal Investigator — First Affiliated Hospital of Fujian Medical University; Minghua Lin, Principal Investigator — Mengchao Hepatobiliary Hospital of Hujian Medical University; Ming Li, Principal Investigator — No.2 People's Hospital of Fuyang City; Xianqiu Huang, Principal Investigator — Guidong People's Hospital of Guangxi Zhuang Autonomous Region; Liying Zhu, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; Lei Yu, Principal Investigator — The Fourth Affiliated Hospital of Harbin Medical University; Baoshan Yang, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Yuguo Zhang, Principal Investigator — The First Hospital of Hebei Medical University; Xiaoli Hu, Principal Investigator — Heilongjiang provincial hospital; Weizhong Yan, Principal Investigator — Jilin Central General Hospital; Xinsheng Xie, Principal Investigator — Affiliated Hospital of Jiaxing University; Caihua Jiang, Principal Investigator — FUJIAN JIANOU HOSPITAL; Guoqi Hu, Principal Investigator — Jieshou City People's Hospital; Junmei Han, Principal Investigator — THE THIRD HOSPITAL OF JIN CHENG; Deshun Yu, Principal Investigator — JIN CHENG PEOPLE'S HOSPITAL; Jianqi Lian, Principal Investigator — Tang-Du Hospital; Jiuping Wang, Principal Investigator — Xijing Hospital; Zhengjun Xu, Principal Investigator — The 910th Hospital; Fenxiang Li, Principal Investigator — LIN FEN THIRD PEOPLE'S HOSPITAL; Tonghe Wu, Principal Investigator — THE SECOND HOSPITAL OF LONGYAN; Fen Wu, Principal Investigator — JIANYANG FIRST HOSPITAL OF NANPING; Yun Wu, Principal Investigator — The Affiliated Hospital of Inner Mongolia Medical University; Houxiong Lin, Principal Investigator — Ningde Municipal Hospital of Ningde Normal University; Yongyue Deng, Principal Investigator — Zhongshan Hospital Xiamen University; Xiao Wang, Principal Investigator — Digestive Diseases Hospital of Shandong First Medical University; Huaizhang Li, Principal Investigator — Shanxi Traditional Chinese Medical Hospital; Liaoyun Zhang, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Binhong Fu, Principal Investigator — Shaowu Municiple Hospital of Fujian Province; Ye Gu, Principal Investigator — The Sixth People's Hospital of Shenyang; Ying Guo, Principal Investigator — The Third People's Hospital of Taiyuan; Ping Li, Principal Investigator — Tianjin Second People's Hospital; Zhifeng Li, Principal Investigator — TONG LIAO INFECTIOUS DISEASES HOSPITAL; Jingning Zhao, Principal Investigator — SINOPHARM TONGMEI GENERAL HOSPITAL; Shuangsuo Dang, Principal Investigator — The Second Affiliated Hospital of Ｘi'an Jiaotong University; Shumei Lin, Principal Investigator — The First Affiliated Hospital of Ｘi'an Jiaotong University; Hongxin Pu, Principal Investigator — Yanbian University Hospital; Li Zhang, Principal Investigator — The Sixth hospital of Handan City; Yongmei Lin, Principal Investigator — Hanzhong 3201 Hospital; Chunzhi Su, Principal Investigator — Hebei Hospital of Traditional Chinese Medicine; Mingxia Jiang, Principal Investigator — Jiamusi Infectious Disease Hospital; Chengrun Xu, Principal Investigator — Southeast Hospital affiliated to Xiamen University; Ying Dai, Principal Investigator — The 7th Hospital of Qiqihar; Jiansheng Huang, Principal Investigator — Wuping County Hospital; Qingrui Peng, Principal Investigator — Xiapu County Hospital; Weixin Wang, Principal Investigator — The 2nd Affiliated Hospital of YCU; Zhigang Lin, Principal Investigator — SanMing Yongan General Hospital; Shihong Wu, Principal Investigator — Yuncheng Central Hospital; Zhongfu Zhao, Principal Investigator — Changzhi Medical College; Yi Zheng, Principal Investigator — Xinhua Hospital of Zhejiang Province
Locations (1):
- Department of Infectious Diseases, The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data would be available to other researchers with the approval of the ethics committee

REFERENCES:
- [Background] Li MH, Xie Y, Zhang L, Lu Y, Shen G, Wu SL, Chang M, Mu CQ, Hu LP, Hua WH, Song SJ, Zhang SF, Cheng J, Xu DZ. Hepatitis B surface antigen clearance in inactive hepatitis B surface antigen carriers treated with peginterferon alfa-2a. World J Hepatol. 2016 May 28;8(15):637-43. doi: 10.4254/wjh.v8.i15.637. PMID 27239256
- [Background] Cao Z, Liu Y, Ma L, Lu J, Jin Y, Ren S, He Z, Shen C, Chen X. A potent hepatitis B surface antigen response in subjects with inactive hepatitis B surface antigen carrier treated with pegylated-interferon alpha. Hepatology. 2017 Oct;66(4):1058-1066. doi: 10.1002/hep.29213. Epub 2017 Aug 26. PMID 28407271
- [Background] Wu F, Lu R, Liu Y, Wang Y, Tian Y, Li Y, Li M, Wang W, Zhang X, Jia X, Dang S. Efficacy and safety of peginterferon alpha monotherapy in Chinese inactive chronic hepatitis B virus carriers. Liver Int. 2021 Sep;41(9):2032-2045. doi: 10.1111/liv.14897. Epub 2021 May 26. PMID 33896094
- [Background] Liu J, Lee MH, Batrla-Utermann R, Jen CL, Iloeje UH, Lu SN, Wang LY, You SL, Hsiao CK, Yang HI, Chen CJ. A predictive scoring system for the seroclearance of HBsAg in HBeAg-seronegative chronic hepatitis B patients with genotype B or C infection. J Hepatol. 2013 May;58(5):853-60. doi: 10.1016/j.jhep.2012.12.006. Epub 2012 Dec 13. PMID 23246508
- [Background] Huang Y, Qi M, Liao C, Xun J, Zou J, Huang H, Long LY, Chen J, Fan X, Chen R. Analysis of the Efficacy and Safety of PEGylated Interferon-alpha2b Treatment in Inactive Hepatitis B Surface Antigen Carriers. Infect Dis Ther. 2021 Dec;10(4):2323-2331. doi: 10.1007/s40121-021-00511-w. Epub 2021 Aug 4. PMID 34350562
- [Background] Zeng QL, Yu ZJ, Shang J, Xu GH, Sun CY, Liu N, Li CX, Lv J, Liu YM, Liang HX, Li ZQ, Pan YJ, Hu QY, Li W, Zhang DW, Wang FS. Short-term Peginterferon-Induced High Functional Cure Rate in Inactive Chronic Hepatitis B Virus Carriers With Low Surface Antigen Levels. Open Forum Infect Dis. 2020 Jun 3;7(6):ofaa208. doi: 10.1093/ofid/ofaa208. eCollection 2020 Jun. PMID 32626791
- [Derived] Chang LJ, Hao CQ, Rao GR, Xu LL, Li J, Cheng Y, Zheng LJ, Wu CW, Chen HX, Chen ZR, Lian JQ, Wu SH, Luo LM, Zhang WL, Zhang Y. Recurrence risk factors for chronic hepatitis B virus-infected patients who achieve functional cure with pegylated interferon-alpha-2b-based therapy: a multicenter pilot study. Virol J. 2025 May 19;22(1):146. doi: 10.1186/s12985-025-02761-3. PMID 40390028